CLINICAL TRIAL: NCT07194681
Title: Regional Nutritional Inequalities and Eating Behaviors Among Turkish Adolescents: A Cross-Regional Analysis
Brief Title: Adolescent Nutrition and Eating Behaviors in Türkiye
Acronym: ANEB-TR
Status: Completed | Type: Observational
Sponsor: Dursun Alper YILMAZ (Other)
Responsible Party: Sponsor-Investigator, Dursun Alper YILMAZ, Res. Asst., Agri Ibrahim Cecen University
Organization: Agri Ibrahim Cecen University (Other)
Other Study IDs: AICU-2025-NUTR01; 112-2025 (Other: Agri Ibrahim Cecen University Ethics Committee)
Record Dates: First submitted 2025-09-19; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Adolescent Nutrition; Eating Behaviors; Nutritional Inequalities; Eating Attitudes
Keywords: Adolescents; Nutrition; Dietary Intake; Eating Attitudes Test (EAT-26); Healthy Nutrition Behavior Scale (HNBS)
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Kırklareli Cohort: Adolescents selected from secondary and high schools in Kırklareli, Türkiye. Observational data collection included 24-hour dietary recall, Healthy Nutrition Behavior Scale (HNBS), and Eating Attitudes Test (EAT-26). No intervention was applied
- Ağrı Cohort: Adolescents selected from secondary and high schools in Ağrı, Türkiye. Observational data collection included 24-hour dietary recall, Healthy Nutrition Behavior Scale (HNBS), and Eating Attitudes Test (EAT-26). No intervention was applied

SUMMARY:
This study examines differences in nutrition and eating behaviors among adolescents living in two regions of Türkiye with contrasting socioeconomic and cultural conditions. A total of 100 adolescents aged 14-18 years were recruited from high schools in Ağrı (Eastern Türkiye) and Kırklareli (Western Türkiye). Participants completed dietary recalls, the Healthy Nutrition Behavior Scale, and the Eating Attitudes Test (EAT-26). The study aims to understand how regional inequalities influence nutrient intake and eating behaviors. Findings may help guide future public health strategies to improve adolescent nutrition across different regions of Türkiye.

DETAILED DESCRIPTION:
Adolescence is a critical developmental stage where nutritional habits are formed and often persist into adulthood. Nutritional inequalities in Türkiye are shaped by socioeconomic and cultural disparities between regions. This cross-sectional observational study was conducted between April and June 2025 in two provinces representing distinct socioeconomic contexts: Ağrı in Eastern Türkiye and Kırklareli in Western Türkiye.

A total of 100 adolescents (50 from each province) aged 14-18 years participated voluntarily. Dietary intake was assessed using 24-hour dietary recalls, and nutrient composition was analyzed with the BeBiS v9.0 software. Healthy eating behaviors were measured with the Healthy Nutrition Behavior Scale (HNBS), and disordered eating attitudes were evaluated with the Eating Attitudes Test (EAT-26).

The primary objective was to compare nutrient intake, healthy eating behaviors, and eating attitudes between the two provinces. Secondary analyses examined whether dietary patterns predicted psychosocial outcomes. Statistical methods included linear mixed-effects models, multivariate analysis of covariance, and principal component regression, adjusting for demographic and socioeconomic covariates.

Ethical approval was obtained from the Ağrı İbrahim Çeçen University Scientific Research and Publication Ethics Committee (Decision No: 112, March 27, 2025). All participants and their guardians provided informed consent.

This study is expected to generate evidence on regional nutritional disparities among adolescents in Türkiye. Results may inform dual public health strategies: (i) improving access to nutrient-dense foods in disadvantaged regions and (ii) addressing over-nutrition and processed food consumption in more affluent regions.

ELIGIBILITY:
Inclusion Criteria:

Adolescents aged 14-18 years

Residing in the study province (Ağrı or Kırklareli) for at least 5 years

Enrolled in selected secondary or high schools

Provided written informed consent (self and parent/guardian)

Exclusion Criteria:

Presence of chronic disease affecting diet (e.g., diabetes, celiac disease)

Currently receiving medical nutrition therapy or weight management interventions

Incomplete dietary recall or questionnaire data

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescents aged 14-18 years attending secondary and high schools in Ağrı (Eastern Türkiye) and Kırklareli (Western Türkiye). Participants were recruited using a two-stage stratified cluster sampling design to reflect urban/rural and school-type diversity.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Eating Attitudes (EAT-26) | Cross-sectional, single assessment (April-June 2025).
  Scores on the Eating Attitudes Test-26 (EAT-26), a validated screening tool for disordered eating attitudes in adolescents
Healthy Nutrition Behavior Score (HNBS) | Single cross-sectional assessment at baseline (April-June 2025).
  Scores on the Healthy Nutrition Behavior Scale (HNBS), a validated 20-item instrument for adolescents. Each item is rated on a 5-point Likert scale (1=never to 5=always). Higher total scores indicate healthier nutrition behaviors.
Nutrient Intake (24-hour recall) | Cross-sectional, single assessment (April-June 2025).
  Energy and nutrient intake (e.g., protein, fat, carbohydrates, vitamins, minerals) based on a 24-hour dietary recall and analyzed using BeBiS v9.0 software.

CONTACTS AND LOCATIONS:
Locations (1):
- Agri Ibrahim Cecen University, Faculty of Health Sciences, Ağrı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study involved a small sample of adolescents, and data include sensitive information on dietary habits and eating attitudes. To protect participant confidentiality, only aggregated results will be published.

REFERENCES:
- [Background] Sezer FE, Alpat Yavas I, Saleki N, Bakirhan H, Pehlivan M. Diet quality and snack preferences of Turkish adolescents in private and public schools. Front Public Health. 2024 Mar 1;12:1365355. doi: 10.3389/fpubh.2024.1365355. eCollection 2024. PMID 38496396
- [Background] Popkin BM, Ng SW. The nutrition transition to a stage of high obesity and noncommunicable disease prevalence dominated by ultra-processed foods is not inevitable. Obes Rev. 2022 Jan;23(1):e13366. doi: 10.1111/obr.13366. Epub 2021 Oct 10. PMID 34632692
- [Background] Neumark-Sztainer D, Wall M, Story M, Fulkerson JA. Are family meal patterns associated with disordered eating behaviors among adolescents? J Adolesc Health. 2004 Nov;35(5):350-9. doi: 10.1016/j.jadohealth.2004.01.004. PMID 15488428
- [Background] Mates E, Lelijveld N, Ali Z, Sadler K, Yarparvar A, Walters T, Brown R, Rodriques B. Nutrition of School-Aged Children and Adolescents in Europe and Central Asia Region: A Literature and Survey Review. Food Nutr Bull. 2023 Mar;44(1):51-61. doi: 10.1177/03795721231163021. Epub 2023 Apr 5. PMID 37017089
- [Background] Aounallah-Skhiri H, Traissac P, El Ati J, Eymard-Duvernay S, Landais E, Achour N, Delpeuch F, Ben Romdhane H, Maire B. Nutrition transition among adolescents of a south-Mediterranean country: dietary patterns, association with socio-economic factors, overweight and blood pressure. A cross-sectional study in Tunisia. Nutr J. 2011 Apr 24;10:38. doi: 10.1186/1475-2891-10-38. PMID 21513570